CLINICAL TRIAL: NCT02405949
Title: GENETIC SUSCEPTIBILITY FACTOR AS A PREDICTOR OF TYPE 2 DIABETES REMISSION AND WEIGHT LOSS AFTER BARIATRIC SURGERY: HOW TO IDENTIFY THE PATIENTS IN WHICH BARIATRIC SURGERY WILL FAIL?
Brief Title: GENETIC SUSCEPTIBILITY FACTOR AS A PREDICTOR OF TYPE 2 DIABETES REMISSION AND WEIGHT LOSS AFTER BARIATRIC SURGERY
Acronym: OBEGEN
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AG) 86/2013
Record Dates: First submitted 2015-03-28; First posted 2015-04-01 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Case-control Study
MeSH Terms: interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- T2D 40%EWL: 15 pacients who had type 2 diabetes before bariatric surgery and presented with less than 40% of the excess weight loss after 12 month from surgery.
  Interventions: Genetic: Genetic test
- nonT2D40%EWL: 15 pacients without type 2 diabetes before bariatric surgery and presented with less than 40% of the excess weight loss after 12 month from surgery.
  Interventions: Genetic: Genetic test
- T2D75%EWL: 35 pacients who had type 2 diabetes befor bariatric surgery and presented with more than 75% of the excess weight loss after 12 month from surgery.
  Interventions: Genetic: Genetic test
- nonT2D75%EWL: 35 pacients without type 2 diabetes befor bariatric surgery and who presented with more than 75% of the excess weight loss after 12 month from surgery.
  Interventions: Genetic: Genetic test

INTERVENTIONS:
Genetic: Genetic test — Analysis of the main genetic variants associated with obesity are evaluated, mainly those related to the regulation of appetite, energy expenditure, adipogenesis, diabetes, inflammation of adipose tissue and others .

SUMMARY:
Obesity is directly related to an increased risk of diabetes mellitus, hypertension, dyslipidemia, cardiovascular disease, and overall mortality. Weight loss is effective in decreasing these risks and to reduce disease severity. Bariatric surgery is an effective therapy for sustained weight loss and type 2 diabetes (T2D) remission in most of the morbidly obese patients. But there is also a significant number of individuals with an inappropriate response to bariatric surgery. Two recent retrospective studies assessed the role of genetic load as a predictor of this response, but the results are still unelucidated. The aim of this study is to assess whether a selection of genetic variants may allow us to identify individuals who will have a satisfactory response after bariatric surgery in terms of weight loss and T2D remission.

DETAILED DESCRIPTION:
A retrospective case-control study of 100 women who underwent bariatric surgery (Roux-en-Y laparoscopic gastric bypass): 50 pacients who were diabetic before surgery: 15 cases with less than 40% of the excess weight loss (EWL) and 35 cases with more than 75% EWL, matched with 50 non diabetic controles: 15 patients with less than 40%EWL and 35 with more than 75%EWL after one year. All individuals were analyzed with a genetic score from Nutri inCode. The predictive ability was analyzed by discrimination (area under the ROC curve), sensitivity and specificity and a score was calculated.

ELIGIBILITY:
Inclusion Criteria:

* women who underwent a gastric bypass with a minimum of 1 year follow-up,
* aged between 18 and 60 years,
* stable weight in the previous 6 months,
* have signed the informed consent.

Exclusion Criteria:

* male,
* with mobility problems that constrain a marked inactivity,
* with pathology that limits the practice of within normal limits (chronic obstructive pulmonary cardiac cerebral vascular-disease, illness, accident sequel, etc ),
* undergoing different surgical techniques to gastric bypass,
* with severe psychiatric disorders or eating disorder.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The trial aimed to recruit a total of 100 female subjects who underwent a gastric bypass in our cente with more than one year of monitoring. These 100 subjects were distributed into 4 subgroups according to the percentage of excess weight loss (%EWL) and the presence or absence of type 2 diabetes before surgery:
  15 women with %EWL <40% without diabetes 15 women with <40%EWL with type 2 diabetes 35 women with a %EWL> 75% without comorbidities 35 women with a %EWL> 75% with type 2 diabetes
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-07; Primary Completion 2013-10 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Predictive value of the genetic test in identifying individuals who will have a good response to bariatric surgery, in terms of weight loss. | 6 month
  Predictive value of the genetic test in identifying individuals who will have a good response to bariatric surgery, in terms of weight loss.
Predictive value of the genetic test in identifying individuals who will have a good response to bariatric surgery, in terms of type 2 diabetes remission after the surgery. | 6 month
  Predictive value of the genetic test in identifying individuals who will have a good response to bariatric surgery, in terms of type 2 diabetes remission.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Vall d´Hebron, Barcelona, Spain